CLINICAL TRIAL: NCT04302051
Title: Feasibility Study for Quantifying Fatty Liver Using Thermo-acoustic Imaging
Brief Title: Assessment of Fatty Liver with Thermo-acoustic Device
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: ENDRA Life Sciences, Inc. (Unknown)
Responsible Party: Principal Investigator, Achuthan Sourianarayanane, Assistant Professor, Medical College of Wisconsin
Other Study IDs: PRO00036361
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: NASH; NAFLD; Non-alcoholic Fatty Liver; Non-Alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis; Fatty Liver; Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Group: The hepatic fat estimation will be performed on the same subjects with the use of the thermo-acoustic device and by MRI-PDFF. The data obtained from the two estimations will be compared.
  Interventions: Diagnostic Test: Thermo-acuostic image acquisition of liver; Diagnostic Test: MRI-PDFF estimation of hepatic fat

INTERVENTIONS:
Diagnostic Test: Thermo-acuostic image acquisition of liver — Estimation of hepatic fat content with thermo-acoustic device
Diagnostic Test: MRI-PDFF estimation of hepatic fat — Estimation of hepatic fat content with MRI

SUMMARY:
The study will evaluate the accuracy of hepatic steatosis estimation by thermo-acoustic ultrasound with estimation by MRI-PDFF (Proton Density Fat Fraction) . It will also evaluate the sensitivity of this device in the diagnosis of fatty liver.

DETAILED DESCRIPTION:
Patients with either known or presumed diagnosis of non-alcoholic fatty liver disease who meets eligibility criteria will be included in the study. They will have imaging done to estimate hepatic steatosis by two modalities (MRI - PDFF and thermo-acoustic ultrasound). The estimation obtained by thermo-acoustic ultrasound will be compared with MRI results for accuracy of estimation by the thermo-acoustic ultrasound device. The study will also evaluate the sensitivity of the thermo-acoustic ultrasound device if it can diagnose the presence of hepatic steatosis when hepatic fat content is 15% or less by volume.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed or suspected to have non-alcoholic fatty liver disease
* Patients 18-70 years of age
* be able to understand and sign on written informed consent
* able to undergo ultrasound and MRI examinations

Exclusion Criteria:

* any metal or electronic implants including but not limited to pacemakers, clips, hips
* known history of pregnancy or becoming pregnant during study period
* unable to understand and sign on written informed consent
* intolerant to ultrasound and/or MRI examinations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult volunteers with diagnosed or suspected for non-alcoholic fatty liver disease will be recruited in the study. Patients who meet inclusion and exclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of hepatic fat estimation by the thermo-acoustic device with MRI-PDFF technique | one year
  The study evaluates if the new thermo-acoustic device can accurately estimate the hepatic fat content among patients with non-alcoholic fatty liver disease to the currently approved method using MRI-PDFF scan.

SECONDARY OUTCOMES:
Evaluate the best and ideal number of the anatomical site for thermo-acoustic evaluation of liver | One year
  The study evaluates the number of estimation required and the appropriate anatomical site to evaluate the liver to obtain best results
Evaluate the sensitivity of the thermo-acoustic device in the diagnosis of hepatic steatosis. | One year
  Evaluate the sensitivity of the thermo-acoustic device in diagnosis presence of hepatic steatosis among patients with MRI-PDFF finding of more than 15% hepatic steatosis

CONTACTS AND LOCATIONS:
Overall Officials: ACHUTHAN SOURIANARAYANANE, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States